CLINICAL TRIAL: NCT04138355
Title: The Clinical Utility of Extracorporeal Shock Wave Therapy on Hand Burns : a Randomized Controlled Study
Brief Title: The Clinical Utility of Extracorporeal Shock Wave Therapy on Hand Burns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hangang Sacred Heart Hospital (Other)
Collaborators: Hallym University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HangangSHH-7
Record Dates: First submitted 2019-10-10; First posted 2019-10-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2019-10

CONDITIONS: Hand Burn
MeSH Terms: interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: The patients' burn scars had re-epithelialized after aseptic care or skin graft. We included patients aged ≥18 years with a deep partial-thickness (second-degree) burn or a full thickness (third-degree) burn to their hands, with joint contracture(hand and wrist), having been transferred to the rehabilitation department after acute burn treatment, and less than 6 months since the onset of the burn injury. Selected patients had a history of hand surgery resulting in painful, retracting scarring on hands.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extracorporeal shock wave therapy group (Experimental): . ESWT was conducted using the Duolith SD-1® device (StorzMedical, Tägerwilen,Switzerland) with an electromagnetic cylindrical coil source for the focused shock wave. ESWT was performed around the primary treatment site at 100 impulses/cm2, an energy flux density(EFD) of 0.05 to 0.30 mJ/mm2, frequency of 4Hz, and 1000 to 2000 impulses were administered at 1-week intervals for 4 sessions.
  Interventions: Other: Extracorporeal shock wave therapy
- conventional manual therapy (No Intervention): the same shock wave equipment used in the experimental group was used with a sham adapter that had the same shape but emitted no energy.

INTERVENTIONS:
Other: Extracorporeal shock wave therapy — ESWT was conducted using the Duolith SD-1® device (StorzMedical, Tägerwilen,Switzerland) with an electromagnetic cylindrical coil source for the focused shock wave. ESWT was performed around the primary treatment site at 100 impulses/cm2, an energy flux density(EFD) of 0.05 to 0.30 mJ/mm2, frequency of 4Hz, and 1000 to 2000 impulses were administered at 1-week intervals for 4 sessions.
  Arms: Extracorporeal shock wave therapy group

SUMMARY:
No study has investigated the effect of extracorporeal shock wave therapy (ESWT) on hand function and hypertrophic scar characteristics. To investigate ESWT effects on burned hands, the investigators compare the results of ESWT combined with manual therapy group to the results of matched conventional(CON) rehabilitation combined with manual therapy group.

DETAILED DESCRIPTION:
Hands are the most frequent injury sites caused by burn, and appropriate rehabilitation is essential to ensure that good functional recovery is achieved. In burn patients, the wound healing process may lead to a fibrotic hypertrophic scar, which is raised, red, inflexible and responsible functional and cosmetic impairments.

This randomized, controlled trial involved 40 patients with burns and dominant right-hand function impairment. Patients were randomized into a ESWT or a CON group. Each intervention was applied to the affected hand for 4 weeks once per week. Hand function was evaluated using the Jebsen-Taylor hand function test (JTT), grasp and pinch power test, and Michigan Hand Outcomes Questionnaire (MHQ). These assessments were evaluated pre-intervention and 4 weeks post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* a deep partial-thickness (second-degree) burn or a full thickness (third-degree) burn to their hands
* less than 6 months since the onset of the burn injury

Exclusion Criteria:

* fourth-degree burns(involving muscles, tendons, and bone injuries)\
* musculoskeletal diseases(fracture, amputation, rheumatoid arthritis, and degenerative joint diseases) in the burned hands
* neurological diseases(such as peripheral nerve disorders)
* preexisting physical and psychologic disability (severe aphasia and cognitive impairment that could influence the intervention)
* severe pain impeding hand rehabilitation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-11-02 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
thickness | 4 weeks
  scar thickness(cm)
melanin and erythema | 4 weeks
  measure melanin levels and the severity of erythema. The higher values indicating a darker and redder skin(AU)
transepithelial water loss | 4 weeks
  the degree of water evaporation
sebum | 4 weeks
  the severity of greese, the higher values indicating a more greese(mg/cm2)
elasticity | 4 weeks
  The numeric values (mm) of the skin's distortion is presented as the elasticity.

SECONDARY OUTCOMES:
grip strength | 4 weeks
  measure grip strength, the higher values indicating a more strength
Jebsen-Taylor hand function test | 4 weeks
  The JTT measure the performance speed of standardized tasks. The JTT involves a series of 7 subtests. We used a scoring system (each subtest score ranged from 0 to 15, and the total score ranged from 0 to 105).

CONTACTS AND LOCATIONS:
Overall Officials: Study Design Participants Intervention Outcome measures Seo, M.D, Study Director — Hangang Scared Heart Hospital
Locations (1):
- Hangang Sacred Heart Hospital, Seoul, Yeong-deungpo-Dong, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] van der Veer WM, Bloemen MC, Ulrich MM, Molema G, van Zuijlen PP, Middelkoop E, Niessen FB. Potential cellular and molecular causes of hypertrophic scar formation. Burns. 2009 Feb;35(1):15-29. doi: 10.1016/j.burns.2008.06.020. Epub 2008 Oct 25. PMID 18952381
- [Result] Cui HS, Hong AR, Kim JB, Yu JH, Cho YS, Joo SY, Seo CH. Extracorporeal Shock Wave Therapy Alters the Expression of Fibrosis-Related Molecules in Fibroblast Derived from Human Hypertrophic Scar. Int J Mol Sci. 2018 Jan 2;19(1):124. doi: 10.3390/ijms19010124. PMID 29301325
- [Result] Cho YS, Joo SY, Cui H, Cho SR, Yim H, Seo CH. Effect of extracorporeal shock wave therapy on scar pain in burn patients: A prospective, randomized, single-blind, placebo-controlled study. Medicine (Baltimore). 2016 Aug;95(32):e4575. doi: 10.1097/MD.0000000000004575. PMID 27512886